CLINICAL TRIAL: NCT00496379
Title: A Phase 2 Study of ZK219477 (ZK-EPO) in Patients With Breast Cancer and Brain Metastases
Brief Title: ZK219477 (Sagopilone) in Patients With Breast Cancer and Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has closed to accrual early due to slow accrual.
Sponsor: Nancy Lin, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Bayer (Industry); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Nancy Lin, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-268
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; CNS Disease
Keywords: metastatic breast cancer; invasive breast cancer; brain metastases; ZK-EPO
MeSH Terms: conditions — Breast Neoplasms; Central Nervous System Diseases; Brain Neoplasms | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZK219477 (Experimental)
  Interventions: Drug: ZK219477

INTERVENTIONS:
Drug: ZK219477 — Given intravenously over approximately 30 minutes once every 3 weeks
  Other Names: ZK-EPO; ZK-Epothilone; Sagopilone

SUMMARY:
The purpose of this research study is to determine the effects (good and bad) of ZK219477(sagopilone) on participants and their cancer. ZK219477 is a chemotherapy drug that is thought to work by interfering with the ability of cancer cells to grow and divide. It is a part of a group of drugs called "epothilones" which appear to cause shrinkage of cancer in some patients with breast cancer. It is generally difficult for chemotherapy to enter the brain. However, it is believed that ZK219477 crosses into the brain. We are also studying whether an investigational MRI scan procedure may eventually help to predict which patients will benefit from ZK219477.

DETAILED DESCRIPTION:
* Participants will be given ZK219477 intravenously over approximately 30 minutes every three weeks.
* During all treatment cycles a physical exam and questions about the participants general health and specific questions about any problems they may be having will be performed.
* At least every three weeks blood tests will be done to assess the effect of ZK219477 on the body.
* After every 2 cycles of treatment, participants will have additional scans to assess the effect of ZK219477 on their cancer. This will include a CT scan of the abdomen, chest, and pelvis, and an MRI of the brain.
* At the time of the standard MRI, participants will be asked to undergo an additional MRI sequence, which means they will be in the MRI machine for approximately 15-20 more minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically invasive breast cancer, with metastatic disease at the time of screening
* Measurable Central Nervous System (CNS) disease, as defined as at least one lesion > or equal too 10mm in longest dimension
* New or progressive CNS lesions after at least one prior standard CNS-directed therapy for treatment of brain metastases, which could include surgical resection, whole brain radiotherapy (WBRT), and/or stereotactic radiosurgery (SRS). Patients must have received prior WBRT, SRS or both.
* Patient has been evaluated by a radiation oncologist, who feels that the plan to evaluate systemic chemotherapy in place of additional brain radiotherapy is an acceptable option
* No increase in corticosteroid use in the week prior to study entry
* Any number prior lines of chemotherapy for metastatic breast cancer
* 18 years of age of older
* Life expectancy of greater than 12 weeks
* ECOG Performance Status 0-2
* Patients must have normal organ function as outlined in the protocol

Exclusion Criteria:

* Patients who have had chemotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients who have had XRT within 3 weeks prior to entering the study or those who have not recovered from adverse events due to XRT
* Patients may not be receiving any other investigational agent
* Patients may not be receiving any cancer-directed therapy
* Prior treatment with investigational chemotherapy for brain metastases
* Prior treatment with epothilone for metastatic breast cancer
* Leptomeningeal carcinomatosis as the only site of CNS involvement.
* Concurrent treatment with an enzyme inducing antiepileptic drug, including phenytoin, carbamezepine, phenobarbital, or oxacarbazepine
* More than 2 seizures over the last four weeks prior to study entry
* Known contraindication to MRI or gadolinium contrast, such as cardiac pacemaker, ocular foreign body, or shrapnel
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at Dana-Farber/Harvard Cancer Center between 8/1/2007-10/29/2009.
Groups:
- Sagopilone: Either 16 mg/m2 or 22 mg/m2 IV Q3W
Period: Overall Study
Arm/Group | Sagopilone
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sagopilone
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate in the Central Nervous System (CNS)
Description: Objective response rate is defined as at least a 50 percent reduction in the Central Nervous system target lesion volume compared to the lesion volume at baseline.
Time Frame: 2 years
Population: The study was closed prior to full accrual as detailed in the manuscript
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sagopilone
Number analyzed (Participants) | 15
percentage of participants | 13.3 [2 to 40]

2. Secondary Outcome: Number of Subjects With Adverse Events (Any Grade)
Description: Adverse events per NCI CTCAE
Time Frame: 2 years
Population: Study was closed prior to full accrual for reasons detailed in published manuscript
Measure: Number; unit: participants
Arm/Group | Sagopilone
Number analyzed (Participants) | 15
participants | 15

3. Secondary Outcome: Objective Response Rate in Non-Central Nervous System (CNS) Sites
Description: Non-CNS response rate (according to RECIST 1.0) limited to patients with measurable non-CNS disease
Time Frame: 2 years
Population: only included the 8 pts with measurable non-CNS disease at baseline. The 7 pts with non-measurable non-CNS disease at baseline were not included in the denominator for this endpoint
Measure: Number; unit: percentage of participants
Arm/Group | Sagopilone
Number analyzed (Participants) | 8
percentage of participants | 0

4. Secondary Outcome: Time to Progression at Any Site.
Description: Time from date of registration until the date of the first documentation of progression or date of death (from any cause),whichever came first, up to 2 years from registration. Progression is defined as either progression in the Central Nervous system (CNS) according to volumetric measurement (Freedman et al. 2011) and /or progression in non-Central Nervous System lesion Measured by RECIST 1.0
Time Frame: 2 years
Population: all patients who received at least 1 dose of protocol therapy
Measure: Median (Full Range); unit: months
Arm/Group | Sagopilone
Number analyzed (Participants) | 15
months | 1.4 [1 to 4]

5. Secondary Outcome: Clinical Benefit Rate.
Description: CBR = CR + PR + SD > 24 weeks in CNS with at least stable non-CNS disease
Time Frame: 2 years
Population: all pts who received at least 1 dose of protocol therapy
Measure: Number; unit: percentage of participants
Arm/Group | Sagopilone
Number analyzed (Participants) | 15
percentage of participants | 13

ADVERSE EVENTS:
Arm/Group | Sagopilone
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sagopilone (N=15)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sagopilone (N=15)
Fatigue (General disorders) | 11 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Neurologic-other (Nervous system disorders) | 1 (1)
Neuropathy-Sensory (Nervous system disorders) | 7 (7)
Dizziness (Nervous system disorders) | 2 (2)
Blurred/Double Vision (Nervous system disorders) | 3 (3)
Eye Pain/ Headache (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Muscle/Joint Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Limb Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 4 (4)
Hypoglycemia (Endocrine disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 1 (1)
Liver Function Tests (Hepatobiliary disorders) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Mucositis (Infections and infestations) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Lymphocytes (Blood and lymphatic system disorders) | 5 (5)
Leukocytes (Blood and lymphatic system disorders) | 3 (3)
Neutrophils (Blood and lymphatic system disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Neuropathy-Motor (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No